CLINICAL TRIAL: NCT02156024
Title: The Short-term Efficacy of Gastrodia and Uncaria Drink in Treating Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Institute of Hypertension (Other)
Responsible Party: Principal Investigator, Cheng Yibang, master, Shanghai Institute of Hypertension
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JDZX2012115
Record Dates: First submitted 2014-05-30; First posted 2014-06-05 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Masked Hypertension
Keywords: clinical trials; Gastrodia and Uncaria Drink
MeSH Terms: conditions — Masked Hypertension | interventions — gastrodin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- placebo (Placebo Comparator): placebo drink, 1 dose at a time, twice a day, duration: 4 weeks
- Gastrodia and Uncaria Drink (Active Comparator): Gastrodia and Uncaria Drink, 1 dose at a time, twice a day, duration: 4 weeks
  Interventions: Drug: Gastrodia and Uncaria Drink

INTERVENTIONS:
Drug: Gastrodia and Uncaria Drink — Gastrodia and Uncaria Drink, 1 dose at a time, twice a day, duration: 4 weeks
  Other Names: tianma gouteng drink
  Arms: Gastrodia and Uncaria Drink

SUMMARY:
The purpose of this study is

1. To determine whether the Gastrodia and Uncaria Drink is effective in the treatment of masked hypertensive patients below 70 years.
2. To find out the suitable groups for the Gastrodia and Uncaria Drink treatment.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 to 70 years
* didn't use any anti-hypertension drugs within 2 weeks
* stage 1 masked hypertensive patients, which means clinic blood pressure<140/90 mmHg,however the daytime(8:00-18:00) 24h ambulatory blood pressure between 135/85 and 150/95mmHg
* be willing to participate in the trials and able to finish clinic visit

Exclusion Criteria:

* secondary hypertension
* be allergic to the clinical trial medicine
* occurrence of stroke, CKD, myocardial infarction within 2 years
* dysfunction of liver or kidney and fundus hemorrhage
* arrhythmia
* ALT, AST, TBL upper the twice of normal range, Scr≥2.0mg/dl, K+≥5.5mmol/L, Urine protein≥2+
* psychiatric disorders
* pregnant, breastfeeding
* other serious conditions in which is not fit for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
blood pressure | March 1,2015

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang DY, Cheng YB, Guo QH, Shan XL, Wei FF, Lu F, Sheng CS, Huang QF, Yang CH, Li Y, Wang JG. Treatment of Masked Hypertension with a Chinese Herbal Formula: A Randomized, Placebo-Controlled Trial. Circulation. 2020 Nov 10;142(19):1821-1830. doi: 10.1161/CIRCULATIONAHA.120.046685. Epub 2020 Oct 6. PMID 33019798
- [Derived] Wei FF, Li Y, Zhang L, Shan XL, Cheng YB, Wang JG, Yang CH, Staessen JA. Persistence of Masked Hypertension in Chinese Patients. Am J Hypertens. 2016 Mar;29(3):326-31. doi: 10.1093/ajh/hpv106. Epub 2015 Jul 6. PMID 26150543